

30.10.2023

# ANKARA MEDIIPOL UNIVERSITY

# Health Sciences Non-Interventional Research Ethics Committee APPLICATION FORM

# 1. DESCRIPTION OF THE RESEARCH

| Title of the Study: | Occupational Eating Disorder in University Students |
|---|---|
| | Effect on Balance |
| <b>English Name of the</b> | The Effect of Eating Disorder on Occupational Balance in |
| Study: | University Students |
| Status of Research: | ( ) Specialization / |
| | Doctoral Thesis ( ) |
| | Master's Thesis |
| | (x) Working for Academic Purposes |
| <b>Nature of the Research:</b> | (x) Questionnaire Survey |
| | () Retrospective Ar Scans Using File and Image Records |
| | ( ) Observational Studies |
| | ( ) Studies with Biochemistry, Microbiology, Pathology and |
| | Radiology Collection Materials such as Blood, Urine, Tissue, |
| | Radiological Images |
| | ( ) Cell and Tissue Culture Studies |
| | () Studies with Materials Obtained During Routine Investigation and |
| | Treatment Procedures |
| | ( ) Studies Based on Anthropometric Measurements and Life |
| | Research on the Evaluation of Habits |
| | ( ) Studies to be Conducted with Genetic Material Excluding Gene |
| | Therapy Clinical Trials and Intended for Identification |
| | () Computerized Test, Interview, Audio/Video Recording |
| | Scientific Researches in which the Data to be Collected will be Used |

#### 2. RESEARCHERS

| | | Title-Name-<br>Surname | Institution/Departm ent | Signature |
|---|---|---|---|---|
| Application | | Lecturer Gör. | Ankara Medipol | |
| | Owne | Büşra KAPLAN | University | |
| r Researcher | | KILIÇ | Occupational<br>Therapy | |
| | | | Department | |

#### 3. INFORMATION ABOUT THE RESEARCH

Purpose and Importance of the Study: It is known that the prevalence of eating disorders is common in university students (1). Eating disorder is defined as a disease that involves less or more food consumption and also leads to physical changes due to mental problems (2). There are also studies that define eating disorder as a psychiatric condition that affects the individual psychosocially, reduces the quality of life and makes it difficult to participate in daily life activities (3). The expression of occupational balance is one of the important concepts determining quality of life, well-being and participation in activities of daily living in occupational therapy discipline (4). This concept varies individually and is related to the amount of occupation, the variety of occupations and the time allocated to occupations during the day (5).

Occupational balance has an important place in affecting the quality of life by enabling individuals to discover the appropriate occupations for themselves and keeping the harmony between these occupations balanced (6,7). When the existing literature is examined, there is no study investigating the effect of eating disorders on occupational balance in our country. With this study, it is aimed to present an original study in the field. In the light of the information obtained from the literature review, it is aimed to examine the effect of eating disorders on occupational balance in university students. Occupation is defined as daily life activities and groups that are named, organized, valuable and meaningful through people and a culture (8).

The aim of this study is to examine the effect of eating disorders on ooccupational balance in university students.

#### Hypotheses

H1: Occupational balance is affected in university students with eating disorders. H1: Occupational balance is affected in university students without eating disorders.

# **Materials and Methods:**

Type of research Cross-sectional study

Population and sample: The population of the study will consist of volunteer students between the ages of 18-25 who are continuing their university education. In the power analysis performed to determine the sample size, it was determined in the G\*Power program, with 95% power (alpha = .05, two-way), the effect size was taken as Cohen's d = 0.5 in accordance with the guidelines provided by J. Cohen, and it was determined that at least 105 people in each group and 210 people in total were needed for the independent sample t-test (9). The result report on the sample test is presented in Appendix 1. Inclusion criteria:

- Volunteering to participate in the study,
- To be able to read and write Turkish,
- 18-25 years of age and studying at undergraduate level Exclusion

#### criteria:

- Having any disability,
- Presence of a chronic disease

Start and end time of the research: November 30, 2023 - August 30, 2024

Forms used in data collection: The individuals included in the study will be evaluated with data collection forms filled in through questionnaires. Demographic information of the individuals (such as class, department, age, gender) will be collected with the sociodemographic information form. Data collection tools will be used by the researchers in face-to-face interviews with the participants and the data will be recorded anonymously.

The data collection tools are;

- 1. Voluntary Consent Form
- 2. Sociodemographic Information Form

Participants who agree to participate in the study and sign the voluntary consent form will be asked to fill in the sociodemographic information form. In the form, information on gender, age, marital status, type of residence, department/grade level studied are questioned.

#### 3. SCOFF Eating Disorders Scale

The Rezzy Eating Disorders Scale will be used to measure whether the participants have an eating disorder. The Turkish validity and reliability of this scale in university students was conducted by Aydemir et al. in 2015. There are five questions in the scale and the questions are answered as yes/no. Yes answer

One point is given for each question answered, and scores of 2 and above are considered as eating disorders (9). This scale will be decisive in the inclusion of the participants in the research and control groups.

### 4. Occupational Balance Questionnaire

The Occupational Balance Questionnaire will be used to measure the occupational balance of individuals. This scale defines the concept of occupational balance by measuring the individual's satisfaction with the number and type of activities of daily living. Each item in the scale is a four-point Likert scale ranging from "strongly agree (0)", "disagree (1)", "agree (2)" and "strongly agree (3)". The scores of all items are summed and written as a total score. Scores that can be obtained in the scale vary between 0-33. A high score is characterized as good occupational balance (10).

It will be determined whether the participants have an eating disorder according to the results of the Rezzy Eating Disorders Scale. Participants with eating disorders will constitute the research group and participants without eating disorders will constitute the control group. Both groups will complete the Occupational Balance Questionnaire and their occupational balances will be compared. The study is planned to be terminated when there are at least 105 participants in each of the research and control groups for the endpoint.

Permissions were obtained for the use of the scales and scale use permissions are presented in Annex-2.

Participants will not be charged and no fee will be paid. Expenses incurred during the reproduction of the questionnaire form will be covered from the budget supported within the scope of TÜBİTAK 2209-A. Informing the participants and obtaining consent that they are volunteers will be carried out by the responsible researcher, Assist. Assist. Büşra Kaplan Kılıç will be the responsible researcher.

**Statistical Method(s):** 'SPSS 20 for Windows' statistical program will be used for statistical analysis. For descriptive data such as sociodemographic information of the participants, frequency and/or mean ± standard deviation (X±SS) values will be used as appropriate. will be given. The data will be examined with normality tests using visual (histogram, probability graphs) and analytical methods (Kolomogrov-Smirnov/ Shapiro-Wilk's test) for the conformity of the data to normal distribution. After the examination, parametric tests will be used if the data are normally distributed and nonparametric tests will be used if the data are not normally distributed.

Statistical significance level will be accepted as p<0.05.

#### **Sources:**

- 1. Kartal, F. T., & Aykut, M. K. (2019). The relationship of social physical anxiety and depression with eating disorder risk in university students. *Journal of Nutrition and Diet*, 47(2), 20-29.
- 2. Patrick, L. (2002). Eating disorders: a review of the literature with emphasis on medical complications and clinical nutrition. (Eating Disorders). *Alternative Medicine Review*, 7(3), 184-203.
- 3. Mahan, L. K., Stump, S. (2008). Krause's Food and Nutrition Theraphy. Saunders Elsevier Publishers, Philadelphia.
- 4. Wagman, P., & Håkansson, C. (2014). Introducing the occupational balance questionnaire (OBQ). *Scandinavian Journal of Occupational Therapy*, 21(3), 227231.
- 5. Yücel, H. (2020). Activity-based occupational therapy. *Hipokrat Bookstore*.
- 6. Wagman, P., Håkansson, C., & Björklund, A. (2012). Occupational balance as used in occupational therapy: A concept analysis. *Scandinavian Journal of Occupational Therapy*, 19(4), 322-327.
- 7. Wagman, P., & Håkansson, C. (2014). Exploring occupational balance in adults in Sweden. *Scandinavian Journal of Occupational Therapy*, 21(6), 415-420.
- 8. Law, M., Polatajko, H., Baptiste, S., & Townsend, E. (1997). Core concepts of occupational therapy. In Canadian Association of Occupational Therapists, Enabling occupation: An occupational therapy perspective (pp. 29-56). *Ottawa, ON: CAOT Publications ACE*.
- 9. Cohen, J. (2013). *Statistical power analysis for the behavioral sciences*. Academic press.
- 10. Aydemir, Ö., Köksal, B., Sapmaz, S. Y., & Yüceyar, H. (2015). Reliability and validity of Turkish form of REZZY Eating Disorders Scale in female university students/Reliability and validity of Turkish form of SCOFF Eating Disorders Scale. *Anatolian Journal of Psychiatry*, 16, 31.
- 11. Günal, A., Pekçetin, S., Demirtürk, F., Şenol, H., Håkansson, C., & Wagman, P. (2020). Validity and reliability of the Turkish occupational balance questionnaire (OBQ11-T). *Scandinavian Journal of Occupational Therapy*, 27(7), 493-499.

#### 4. INFORMED CONSENT FORM

#### Dear Participant

- 1. This study you are participating in is a research titled "The Effect of Eating Disorder on Occupational Balance in University Students".
- 2. The aim of the study was to investigate the effects of disordered eating on occupational balance in university students.
- **3.** The study will be conducted with 210 volunteer participants who are studying at Ankara Medipol University, meet the inclusion criteria and agree to be included in the study.
- **4.** During the research, data will be collected face-to-face with the survey method using the Rezzy Eating Disorders Scale and the Occupational Balance Questionnaire.
- **5.** If you participate in the survey, you will be asked to fill in the questionnaire forms in approximately 10-15 minutes.
- **6.** There is no risk to which you will be exposed.
- 7. With the data to be obtained, it is aimed to examine the effects of university eating disorder on ooccupational balance. The results of our study will help us to make various suggestions to reduce the negative conditions caused by eating disorders.
- **8.** There are no alternative methods or treatment schemes that can be applied to you and their possible benefits and risks.
- 9. No compensation or treatment of any kind will be provided to you.
- 10. You will not be reimbursed for expenses such as transportation and meals.
- 11. Your participation in this research is entirely voluntary and you may refuse to participate or withdraw from the research at any time, without any penalty or sanction and without losing any rights.
- 12. The data collected from you may be directly accessible to monitors, surveyors, ethics committees, institutions and other relevant health authorities, but this information will be kept confidential. By signing the written informed consent form, you consent to such access by the subject or his/her legal representative.
- 13. In accordance with the relevant legislation, the records that will reveal the identity of the volunteer will be kept confidential and cannot be disclosed to the public; even if the research results are published, the identity of the volunteer will remain confidential.
- **14.** You will be informed in good time when new information becomes available that is relevant to the research topic and may affect your willingness to continue to participate in the research.

- **15.** To provide more information about the research, your own rights, or any adverse events related to the research, you can contact the Research Assistant. Prof. Dr. Büşra KAPLAN KILIÇ at 05543303227 24 hours a day.
- **16.** At any stage of the research, if you do not wish to participate in the research, you can withdraw from the research.
- 17. The estimated time to continue the research is 10-15 minutes.
- **18.** The estimated number of volunteers expected to participate in the research is 210.
- 19. No biological material will be obtained from you.

# 20. (Participant's Declaration)

"I have read all the explanations in the Informed Voluntary Consent Form. I have been given a written and verbal explanation about the research, the subject and purpose of which are stated above, by the physician named below. I understand that I am participating in the research voluntarily and that I can withdraw from the research at any time with or without reason."

- 21. "I agree to participate in this research voluntarily, without any pressure or coercion."
- 22. Volunteer

Name/surname/signature/date

- 23. Principal Investigator Lecturer. Assist. Büşra KAPLAN KILIÇ
- 24. Witness:

Name/surname/signature/date

- 25. No legal representative is needed.
- 26. There is no genetic research on biological material obtained from volunteers.